CLINICAL TRIAL: NCT01305330
Title: Role of Active Surveillance and Identification of Prognostic Factors for Progression in Early Stage Renal Cell Carcinoma
Brief Title: The Natural History of Small Renal Masses
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Kidney Foundation of Canada (Other); Canadian Urologic Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: SRM
Record Dates: First submitted 2011-02-18; First posted 2011-02-28 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Patients With Newly Diagnosed Small Renal Masses(<4cm)
Keywords: small renal mass; active surveillance; kidney mass; kidney tumour
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsy cores, nephrectomy tissue, and blood and urine will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is a rising incidence of incidentally detected small renal tumours due to improved imaging techniques. Traditionally, patients diagnosed with these small renal masses undergo surgery and therefore there is limited data about the natural history of these tumours. Several small series have reported that most of these small masses grow slowly and might not require early intervention and that only some masses grow rapidly requiring immediate surgery. Presently, the investigators have not been able to identify prospectively which masses are going to grow slowly. The investigators plan to use computed tomography (CT) and Magnetic Resonance Imaging (MRI) parameters, microsatellite analysis and tissue analysis to determine which masses will behave more aggressively. Additionally, the observations on the natural history of small renal masses need to be validated with a multicentric and systematically followed cohort.

DETAILED DESCRIPTION:
Hypothesis

Since most renal cell carcinomas (RCC's) that are now detected by imaging as small renal masses, grow slowly and remain asymptomatic for years, we hypothesize that:

* Small RCC's that are destined to metastasize do so early or after they reach a larger size
* Delayed surgical treatment of asymptomatic, incidentally detected, small RCC's WILL NOT have a significant impact on overall survival
* The majority of small RCC's MAY NOT need to be treated.
* RCC's that are destined to progress can be identified by abnormal perfusion patterns on imaging and by their cellular and genomic characteristics on needle biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic T1a (< 4.0 cm) renal mass and unfit for surgery due to advanced age or co-morbidity, OR
* Asymptomatic T1a (< 4.0 cm) and refusal of surgery
* No evidence of metastatic disease (N0M0)
* Preparedness to comply with a close follow-up protocol
* Informed consent

Exclusion Criteria:

* Life expectancy < 2 years
* Already being followed for a small renal mass for more than 12 months
* Concurrent systemic therapy for other malignancies
* Known hereditary renal cancer syndromes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2004-08; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Tumour progression: | 4 times year 1, 2 times year 2 and 3, yearly thereafter
  i) calculated tumour volume doubles (100% increase) within any one-year period, and/or ii) the maximum tumour diameter reaches 4 cm., and/or iii) patients develop symptoms considered to be possibly due to their renal tumour and/or iv) patients develop metastases

SECONDARY OUTCOMES:
Time to Tumour Progression | 4 times year 1, 2 times year 2 and 3, yearly thereafter
  Time to tumour progression will be measured from the date of diagnosis to the date of progression or, if progression has not occurred, until the date of last follow-up.
Growth rate | 4 times year 1, 2 times year 2 and 3, yearly thereafter
  Defined by volume (cm3 ) measured over time (years). Tumour bi-dimensional diameter will be recorded and reported to allow comparison with the literature to date. Tumour volume will be calculated from follow-up images using the formula for ellipsoid volume: 0.5326 x X x Y x Z.

CONTACTS AND LOCATIONS:
Overall Officials: Michael AS Jewett, MD, FRCSC, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- Princess Margaret Hospital, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No